CLINICAL TRIAL: NCT00066183
Title: Studies in Phosphorus Metabolism
Brief Title: Studying Phosphorus Metabolism
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030254; 03-D-0254
Record Dates: First submitted 2003-08-04; First posted 2003-08-05 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-01

CONDITIONS: Phosphorus Metabolism
Keywords: Fibroblast Growth Factor 23; FGF-23; Hypophosphatemia; Phosphaturia; Phosphorus; Phosphorus Metabolism
MeSH Terms: conditions — Hypophosphatemia; Hypophosphatemia, Familial

SUMMARY:
Phosphorus and phosphate irons play critical roles in bone structure and essential cellular functions.

The purpose of this study is to learn more about the factors and hormones that regulate phosphorus in the body by collecting blood and urine samples from patients with disorders of phosphate control.

Both children and adults will be enrolled in this study. Researchers will collect blood and urine samples from participants on multiple occasions (2 to 6 times). Some blood specimens will be taken after an overnight fast and participants may be asked to collect all their urine during a 24-hour period. Researchers will analyze these blood and urine samples to better understanding how the body handles phosphorus.

DETAILED DESCRIPTION:
Phosphorus and phosphate ions play an important role in cellular metabolism as well as bone structure. Scientific evidence suggests that, in addition to Vitamin D and PTH systems, novel factors, such as Fibroblast Growth Factor 23 (FGF-23) and Matrix extracellular phosphoglycoprotein (MEPE), may play an important role in phosphorus regulation. These factors have been best studied in rare genetic and acquired phosphate wasting disorders such as tumor induced osteomalacia (TIO), X linked hypophosphatemia (XLH) and autosomal dominant hypophosphatemic rickets (ADHR). Patients with other abnormal phosphate regulating states such as hyperparathyroidism and hypoparathyroidism, pseudohypoparathyroidism etc. undergoing phosphorus-altering interventions may provide important insight into the role of these hormones.

We are proposing an observational study with collection of blood and urine samples to study both established (e.g. mineral ions, bone markers, PTH-Vit D system, TMP-GFR) and novel (e.g. FGF-23 and MEPE) constituents of the phosphorus metabolism pathway. Patients with abnormal phosphorus regulating states will be enrolled and we will study the natural history of their disease and the effects of specific interventions that are likely to change phosphorus balance.

The outcome will potentially aid understanding of this new field of mineral regulating hormones and generate both interest and research in phosphorus metabolism. It is hoped that this will also encourage clinical trials in treatment of phosphate wasting disorders.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients of any age, gender or ethnicity who will help fulfill the objectives laid out in Section II.

We propose to study patients primarily enrolled in other clinical center protocol(s). They will continue to receive treatment/ interventions per the original protocols.

EXCLUSION CRITERIA:

Patients with significant cognitive impairment who are unable to give informed consent or patients having other significant mineral disturbances that could confound the parameters being studied will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2003-08; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Murer H, Forster I, Hernando N, Lambert G, Traebert M, Biber J. Posttranscriptional regulation of the proximal tubule NaPi-II transporter in response to PTH and dietary P(i). Am J Physiol. 1999 Nov;277(5):F676-84. doi: 10.1152/ajprenal.1999.277.5.F676. PMID 10564230
- [Background] Cai Q, Hodgson SF, Kao PC, Lennon VA, Klee GG, Zinsmiester AR, Kumar R. Brief report: inhibition of renal phosphate transport by a tumor product in a patient with oncogenic osteomalacia. N Engl J Med. 1994 Jun 9;330(23):1645-9. doi: 10.1056/NEJM199406093302304. No abstract available. PMID 8177270
- [Background] Jonsson KB, Mannstadt M, Miyauchi A, Yang IM, Stein G, Ljunggren O, Juppner H. Extracts from tumors causing oncogenic osteomalacia inhibit phosphate uptake in opossum kidney cells. J Endocrinol. 2001 Jun;169(3):613-20. doi: 10.1677/joe.0.1690613. PMID 11375132